CLINICAL TRIAL: NCT04421391
Title: Phase II Study of QuadraMune(TM) for Prevention of COVID-19 in High Risk Populations
Brief Title: QuadraMune(TM) for Prevention of COVID-19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Therapeutic Solutions International (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QuadraMune002
Record Dates: First submitted 2020-06-04; First posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Covid19; Coronavirus; SARS-CoV 2
Keywords: Immunology; Innate Immune System
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): Patients will receive 2 pills of QuadraMune(TM) daily for 12 weeks
  Interventions: Dietary Supplement: QuadraMune(TM)

INTERVENTIONS:
Dietary Supplement: QuadraMune(TM) — QuadraMune(TM) is a commercially available nutritional supplement

SUMMARY:
QuadraMune(TM) is a nutritional supplement which has previously been demonstrated to possess antiinflammatory and immune modulatory activity based on in vitro and pilot in vivo studies. The current clinical trial aims to assess in a 500 volunteer trial the efficacy of QuadraMune(TM) in reducing infection in individuals at high risk of COVID-19.

DETAILED DESCRIPTION:
QuadraMune(TM) is composed of 4 natural ingredients.

Pterostilbene is an analogue of resveratrol, and has been shown to possess antiinflammatory activity. Additionally, this compound suppresses macrophage activation while enhancing NK activity.

Epigallocatechin gallate (EGCG) is one of the active ingredients in green tea and has been shown to act as an activator of T cells, and a suppressor of neutrophil mediated inflammation.

Sulforaphane is derived from broccoli and studies have shown that it protects lungs from inflammatory pathology.

Thymoquinone, which is chemically related to hydroxychloroquine, possessing antiviral effects and increases NK activity.

QuadraMune is a combination of these ingredients and is believed to possess superior in vitro and in vivo therapeutic properties as compared to when the ingredients are administered individually.

The study aims to assess preventative effects of QuadraMune(TM) administration for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent, provided electronically via the EDC, demonstrating the subject understands the procedures required for the study and the purpose of the study Male or female patients 18 years of age or older that are considered to be high-risk individuals.
* High-risk individuals are defined as all health care workers in hospitals, clinics, and emergency rooms, and medical facilities.
* Subjects must agree to practice at least two highly effective methods of birth control for the duration of the study This includes condoms with spermicide, oral birth control pills, contraceptive implants, intra-uterine devices, or diaphragms. At least one of these must be a barrier method. Subjects not of reproductive potential will be exempt (e.g. post-menopausal, surgically sterilized)

Exclusion Criteria:

* Refusal to provide informed consent Any previous positive test for COVID-19 by RT-PCR Symptomatic for COVID-19 Diarrhea prior to the start of treatment Type I or II diabetes Atherosclerotic Coronary Artery Disease

Any contraindication for treatment with hydroxychloroquine including:

Hypoglycemia G6PD deficiency Porphyria Anemia Neutropenia Alcoholism Myasthenia Gravis Skeletal muscle disorder Maculopathy Changes in the visual field Liver disease, with ALT/AST > 2.5 upper limit normal and total bilirubin >2.5 upper limit normal Psoriasis Any comorbidities which, in the opinion of the investigator, constitute health risk for the subject.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2020-06-08 (Estimated); Primary Completion 2020-11-01 (Estimated); Study Completion 2020-11-08 (Estimated)

PRIMARY OUTCOMES:
Prevention of COVID-19 | 12 Weeks
  Prevention of COVID-19 symptoms as recorded in a daily diary

SECONDARY OUTCOMES:
Safety as determined by presence or absence of Adverse Events and Serious Adverse Events | 12 Weeks
  Assessment of adverse events and serious adverse events will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: James Veltmeyer, MD, Principal Investigator — Therapeutic Solutions International
Locations (1):
- Therapeutic Solutions International, Oceanside, California, United States

IPD SHARING:
Plan to Share IPD: Undecided